CLINICAL TRIAL: NCT01515254
Title: The Feeding Dynamic Intervention Study
Brief Title: The Feeding Dynamic Intervention: Self Regulation of Intake in Preschoolers
Acronym: FeeDIn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ihuoma Eneli, Medical Director, Center for Healthy Weight and Nutrition; Professor of Pediatrics, The Ohio State University, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB11-00399; 1R03DK089198-01A1 (NIH)
Record Dates: First submitted 2012-01-18; First posted 2012-01-24 (Estimated); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Children; Exogenous Obesity; Eating Behavior
Keywords: Children; Obesity Prevention; Child Overweight; Energy Compensation; Eating Behavior; Food Intake; Parenting Behavior
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No intervention- control group (No Intervention): Visits to physicians, WIC offices, nutrition program etc will be tracked. The subjects will undergo the energy regulation tests at baseline and 3 months. They will complete surveys and have their weight taken. The control group subjects will have the opportunity to receive the intervention at the end of the study
- lifestyle counseling, parental feeding (Experimental): Intervention group subjects will undergo a Feeding Dynamic Intervention (FDI). The intervention will be delivered in a closed group setting and will consist of 6 intervention sessions lasting 90 minutes each. Visits to physicians, WIC offices, nutrition program etc will be tracked. The subjects will undergo the energy regulation tests at baseline and 3 months. They will complete surveys and have their weight taken.
  Interventions: Behavioral: lifestyle counseling, parental feeding

INTERVENTIONS:
Behavioral: lifestyle counseling, parental feeding — Intervention group subjects will undergo a Feeding Dynamic Intervention (FDI). The intervention will be delivered in a closed group setting and will consist of 6 intervention sessions lasting 90 minutes each. Visits to physicians, WIC offices, nutrition program etc will be tracked. The subjects will undergo the energy regulation tests at baseline and 3 months. They will complete surveys and have their weight taken.
  Arms: lifestyle counseling, parental feeding

SUMMARY:
In this study the investigators will examine the Feeding Dynamic Intervention (FDI) as a tool to prevent obesity in young children. The purpose of the intervention is to improving caregiver feeding practices, child eating behaviors, and child self-regulation of energy intake in the short term.

DETAILED DESCRIPTION:
Childhood obesity is a significant public health problem. In the last three decade, there has been a marked increase in the prevalence of childhood obesity. Currently, 23% of preschoolers (2-5 years) in the United States are overweight or obese, a critical period to target in hopes of reversing this trend. The purpose of this study is to test the efficacy of a novel obesity intervention program for preschool-aged children. Emerging consensus indicates that excessive, intrusive, overt control in feeding or a chaotic non-structured feeding environment are risk factors for childhood obesity. The 2007 Expert Committee Recommendations on the Prevention, Assessment, and Treatment of Childhood Obesity specifically identified maternal feeding practices as important, categorically stating there is consistent evidence to support "avoiding overly restrictive feeding behaviors." The guidelines emerged from a growing body of literature indicating that overly controlling caregiver feeding behaviors, in particular, significantly increase children's obesity risk.

Despite the evidence for the importance of feeding dynamics, no childhood obesity interventions focused on this area have been rigorously tested. The Feeding Dynamic Intervention (FDI) is a 12-week educational intervention. The intervention will be delivered in a closed group setting and will consist of 6 intervention sessions lasting 90 minutes each. We will recruit 84 mothers with 3- to 5-year-old obese children, randomly assigned to either the FDI or a comparison to a waiting list control group (WLG). At the end of the 6 month study we will assess knowledge and behavioral changes between the groups on (i) maternal self-reported feeding practices; (ii) improving energy compensation (COMPX), decreasing Eating in the Absence of Hunger (EAH) and increasing mother-reported satiety responsiveness in their child. Finally, we will investigate an exploratory hypothesis that children in the FDI group, compared to children in the wait-list control group, will demonstrate a lower increase in body mass index (BMI) z-score over 6 months.

ELIGIBILITY:
Inclusion Criteria:

* The child is between ages 3-5 years (36 to 71 months). [Note if a family has more than one qualifying child we will choose the child with the lower CEBQ SR score and if they are equal we will randomly select the target child for the study dyad.]
* Child's body mass index > 85th percentile for age and sex
* This will be calculated based on age, weight and height using the Center for Healthy Weight and Nutrition BMI calculator [if mother is unsure of the weight and height ask whether she has been told her child is overweight or obese by the PCP]
* Child has significantly abnormal parent-reported impairment of energy regulation (Rating of 2.8 or lower on the CEB-Q).
* The mother is fluent in English (measures are limited to English at this time)
* Mother (or female caregiver) has primary legal and physical custody of the child and is primarily responsible for feeding the child. Specifically the child is not in a non-parental home daycare more than 20 hours/week. Structured child care centers are not included in this limitation because they use structure care and feeding techniques similar to those taught in the FeeDIn Program.

Exclusion Criteria:

* Child has a medical condition or takes a medication that affects appetite, eating, or growth;
* Child has food allergies or dietary restrictions that interfere with feeding or the study tests (i.e., milk, gluten and eggs?)
* Child has any developmental or behavioral diagnosis that might affect his/her ability to respond to a behaviorally-based intervention, e.g., cognitive impairment, language delay, or autism.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2012-02; Primary Completion 2018-06 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Increased Energy Regulation | Change from baseline in energy compensation at 3 months and Change from baseline in energy compensation at 6 months
  Children in the FDI group, compared to children in the wait-list control group will show improved energy compensation regulation (COMPX), decreased Eating in the Absence of Hunger (EAH), and increasing Satiety Responsiveness (CEBQ-SR).

SECONDARY OUTCOMES:
Reduce BMI | Change from baseline in BMI-z score at 3 months and Change from baseline in BMI-z score at 6 months
  Children in the FDI group, compared to children in the wait-list control group, will demonstrate a lower increase in body mass index (BMI) z-score over 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ihuoma Eneli, MD, MS, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Eneli IU, Tylka TL, Hummel J, Watowicz RP, Perez SA, Kaciroti N, Lumeng JC. Rationale and design of the Feeding Dynamic Intervention (FDI) study for self-regulation of energy intake in preschoolers. Contemp Clin Trials. 2015 Mar;41:325-34. doi: 10.1016/j.cct.2015.01.006. Epub 2015 Jan 20. PMID 25616192